CLINICAL TRIAL: NCT06439043
Title: Developing a Culturally and Methodologically Adapted EMDR Protocol for the Treatment of Major Depressive Disorder and Determining Its Efficacy by Testing it Through Online and Face-to-face Modes of EMDR Therapy
Brief Title: Cultural Adaptation of EMDR for Major Depressive Disorder and Compaire Its Online and Face-to-Face Testing
Acronym: EMDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khushal Khan Khattak Univeristy, Karak, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Anwar Khan, PhD Student, University Malaysia Sarawak
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1213
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder 1
Keywords: Depressive Disorder, Major
MeSH Terms: conditions — Major Depressive Disorder 1; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The adapted EMDR treatment protocol will be administered both online and face-to-face. Patients will be randomly allocated to either the face-to-face mode or the online mode of EMDR at the same time.
Who Masked: Participant
Masking Description: It will be a single-blinded study in which only the participants will be unaware of certain aspects of the research design. Typically, this means that the participants will not know which treatment they are receiving or the mode of treatment (online or face-to-face), while the researchers administering the treatment and collecting data will be aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face to Face Eye Movement Desensitization & Reprocessing Therapy (Experimental): The face-to-face Eye Movement Desensitization and Reprocessing (EMDR) therapy will be administered by the psychotherapist at their clinic. The treatment will consist of a total of 12 to 13 sessions, with one session conducted per week.
  Interventions: Other: EMDR Psychotherapy
- Online Eye Movement Desensitization and Reprocessing therapy (Active Comparator): The online Eye Movement Desensitization and Reprocessing (EMDR) therapy will be administered by the psychotherapist using BilateralBase software. The treatment will consist of 12 to 13 online sessions, with one session conducted per week.
  Interventions: Other: Online EMDR Psychotherapy

INTERVENTIONS:
Other: EMDR Psychotherapy — EMDR psychotherapy will be delivered in person by the psychotherapist to treat symptoms of Major Depressive Disorder, consisting of 12 weekly sessions.
  Arms: Face to Face Eye Movement Desensitization & Reprocessing Therapy
Other: Online EMDR Psychotherapy — Online EMDR Psychotherapy will be delivered online by the psychotherapist to treat symptoms of Major Depressive Disorder, consisting of 12 weekly sessions.
  Arms: Online Eye Movement Desensitization and Reprocessing therapy

SUMMARY:
The present study aims to develop a culturally and methodologically adapted EMDR therapy protocol, determine its treatment fidelity, and then clinically test its efficacy in the treatment of Major Depressive Disorder in Pakistan by utilizing both in-person and online modalities of EMDR therapy.

DETAILED DESCRIPTION:
Background and Aim: Major Depressive Disorder(MDD) is a globally leading cause of disability. Currently, psychotherapies like Eye Movement Desensitization and Reprocessing(EMDR) and Cognitive Behavioral Therapy(CBT) are widely available. Since EMDR originated in the United States, it may not be completely appropriate for non-Western countries like Pakistan, necessitating possible modifications. Moreover, therapists have long practiced face-to-face EMDR, but recently, online EMDR modalities have emerged. Nonetheless, it is surprising that there is a dearth of research not only on adaptations of EMDR in Pakistan but also on testing its clinical efficacy, particularly its online modalities. Considering this, the present study aims to develop a culturally and methodologically adapted EMDR therapy protocol, and clinically evaluate its efficacy in treating MDD in Pakistan by comparatively administering it through in-person and online modalities. Methods: This study will employ a mixed mode Randomized Controlled Trial design with a consecutive sample of (n=90). Patients will be treated by using adapted EMDR therapy protocol. Patients will be randomly allocated to in-person and online modes of EMDR. Various qualitative methods and quantitative techniques will be employed to data. Conclusion: This study is likely to make significant contributions by delivering insights about how to develop culturally and methodologically adapted EMDR. This study will extend our knowledge about the comparative effectiveness of EMDR in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should exhibit symptoms of Major Depressive Disorder.
2. Male and female patients will be chosen equally.
3. Patients between the ages of 20 and 50 will be selected.
4. Patients should preferable be "treatment-naïve," meaning they have no recent history of any psychotherapy or medication.

Exclusion Criteria:

a. There must be no significant neuropsychological or cognitive disorders among the patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — both male and female patients will be selected
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Major Depressive Disorder | 6 months
  Major Depressive Disorder will be assess by Hamilton Depression rating scale with score more than 30 as cut off point

CONTACTS AND LOCATIONS:
Locations (1):
- KKKUk, Kohat, Pakistan